CLINICAL TRIAL: NCT06849128
Title: Effects of NeuroReAlign Therapy on Cognition in Patients with Stroke: a Randomized Controlled Trial
Brief Title: NeuroReAlign Therapy for Cognitive Rehabilitation in Patients with Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Anas Radi Hassan Alashram, Assistant Professor, Middle East University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ADA/1100
Record Dates: First submitted 2025-02-20; First posted 2025-02-27 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional cognitive training (Active Comparator): A conventional cognitive training protocol involves structured, repetitive exercises designed to enhance specific cognitive functions, such as memory, attention, executive function, and processing speed. These training programs are delivered through paper-and-pencil tasks, computer-based exercises, and therapist-guided activities. Tasks used include working memory exercises (e.g., digit span recall), attention training (e.g., Stroop test, visual scanning), problem-solving activities (e.g., Tower of Hanoi), and language exercises (e.g., verbal fluency tasks), for 45 minutes per session, 3 times weekly, for 4 weeks.
  Interventions: Other: Conventional cognitive training
- NeuroReAlign Therapy (Experimental): Patients in this group will receive NeuroReAlign Therapy, including motor training (e.g., treadmill training, balance training), multimodal sensory stimulation (e.g., proprioceptive and visual), cognitive training (e.g., traditional cognitive exercise), and motivation, for 45 minutes per session, 3 times weekly, for 4 weeks.
  Interventions: Other: NeuroReAlign Therapy

INTERVENTIONS:
Other: NeuroReAlign Therapy — Patients in this group will receive NeuroReAlign Therapy, including motor training (e.g., treadmill training, balance training), multimodal sensory stimulation (e.g., proprioceptive and visual), cognitive training (e.g., traditional cognitive exercise), and motivation, for 45 minutes per session, 3 times weekly, for 4 weeks.
  Arms: NeuroReAlign Therapy
Other: Conventional cognitive training — A conventional cognitive training protocol involves structured, repetitive exercises designed to enhance specific cognitive functions, such as memory, attention, executive function, and processing speed. These training programs are delivered through paper-and-pencil tasks, computer-based exercises, and therapist-guided activities. Tasks used include working memory exercises (e.g., digit span recall), attention training (e.g., Stroop test, visual scanning), problem-solving activities (e.g., Tower of Hanoi), and language exercises (e.g., verbal fluency tasks), for 45 minutes per session, 3 times weekly, for 4 weeks.
  Arms: Conventional cognitive training

SUMMARY:
The goal of this randomized controlled trial is to investigate the effects of NeuroReAlign Therapy on cognition in stroke survivors in the chronic stage (>6 months). The study will include male and female participants aged 18-70 years.

The main questions it aims to answer are:

Does NeuroReAlign Therapy improve cognition in stroke survivors compared to conventional physiotherapy? Researchers will compare NeuroReAlign Therapy to conventional cognitive therapy to determine its effects on cognition.

Participants will:

Undergo NeuroReAlign Therapy or conventional cognitive therapy for 4 weeks. Have their cognition evaluated using the Montreal Cognitive Assessment (MoCA), Mini-Mental State Examination (MMSE), Trail Making Test (TMT), Stroop Test, Digit Span Test, and Verbal Fluency Test (VFT).

Complete outcome assessments at baseline and after the intervention (week 4).

ELIGIBILITY:
Inclusion Criteria:

* Patients with ischemic or hemorrhagic stroke
* Have a stroke more than 6 months
* Age between 18 and 70

Exclusion Criteria:

* Patients with severe cognitive impairments
* Patients cannot walk independently

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-04-15 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | At baseline (week 0) and post-intervention (week 4)
  The Montreal Cognitive Assessment (MoCA) is a widely used screening tool designed to assess mild cognitive impairment in stroke survivors and other neurological populations. It evaluates multiple cognitive domains, including attention, memory, visuospatial abilities, executive function, language, and orientation. The test consists of 30 points, with a cutoff score of <26 suggesting cognitive impairment. The MoCA is sensitive to subtle cognitive deficits and is particularly useful in detecting post-stroke cognitive impairments that may not be captured by other general cognitive tests.

SECONDARY OUTCOMES:
Mini-Mental State Examination (MMSE) | At baseline (week 0) and post-intervention (week 4)
  The Mini-Mental State Examination (MMSE) is a brief, standardized cognitive test used to assess overall cognitive function in stroke survivors. It evaluates orientation, attention, memory, language, and visuospatial skills, with a total score of 30 points. Lower scores indicate greater cognitive impairment, with a cutoff of ≤24 typically suggesting cognitive dysfunction. Although widely used, the MMSE may be less sensitive to detecting mild cognitive impairment compared to the Montreal Cognitive Assessment (MoCA).
Trail Making Test (TMT) | At baseline (week 0) and post-intervention (week 4)
  The Trail Making Test (TMT) is a neuropsychological test used to assess processing speed, attention, and executive function in stroke survivors. It consists of two parts: TMT part A, where participants connect numbers in ascending order to measure processing speed and visual search, and TMT part B, where they alternate between numbers and letters (1-A-2-B, etc.) to assess cognitive flexibility and executive function. Longer completion times indicate greater impairment. The TMT is widely used to evaluate cognitive deficits following stroke, particularly in domains related to attention and task-switching.
Stroop Test | At baseline (week 0) and post-intervention (week 4)
  The Stroop Test assesses cognitive control, attention, and response inhibition, which are often affected after a stroke. It requires participants to name the color of printed words while ignoring the actual word meaning (e.g., saying "blue" when the word "RED" is printed in blue ink). The test measures processing speed, selective attention, and executive function by evaluating the ability to suppress automatic responses. Poor performance on the Stroop Test may indicate deficits in cognitive control and attention regulation, which are common in post-stroke cognitive impairment.
Digit Span Test | At baseline (week 0) and post-intervention (week 4)
  The Digit Span Test, a subtest of the Wechsler Adult Intelligence Scale (WAIS), assesses attention, working memory, and verbal short-term memory. Participants are asked to repeat a series of numbers in the same order (forward digit span) or in reverse order (backward digit span). The backward span is particularly sensitive to working memory deficits, which are frequently observed in stroke survivors. This test is simple yet effective in evaluating short-term memory and cognitive processing capacity.
Verbal Fluency Test (VFT) | At baseline (week 0) and post-intervention (week 4)
  The Verbal Fluency Test (VFT) measures language function, executive control, and processing speed. It consists of two types: phonemic fluency, where participants generate words starting with a specific letter, and semantic fluency, where they list words within a given category (e.g., animals). The number of correct words generated within a time limit (usually 60 seconds) reflects cognitive function, with lower scores indicating language or executive dysfunction. This test is commonly used to assess cognitive deficits in post-stroke patients, particularly those affecting language and retrieval ability.